CLINICAL TRIAL: NCT06882343
Title: Performance of Bioactive Low Viscosity Composite in Deep Marginal Elevation Restorations: a Randomized Clinical Trial
Brief Title: Performance of Bioactive Low Viscosity Composite in Deep Marginal Elevation Restorations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Hossam Elmoaty, Dentisy, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ahmed elmoety protocol
Record Dates: First submitted 2025-03-08; First posted 2025-03-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Deep Caries; Caries, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bioactive Giomer Material (Active Comparator)
  Interventions: Other: Beautiful Flow Plus X
- Nanohybrid resin composite (Active Comparator)
  Interventions: Other: Dentsply Nanohybrid flowable composite

INTERVENTIONS:
Other: Beautiful Flow Plus X — Shofu's Beautifil Flow Plus X F03 is an advanced injectable bioactive composite that merges the adaptability of flowable composites with the mechanical properties of hybrid composites
  Arms: Bioactive Giomer Material
Other: Dentsply Nanohybrid flowable composite — a conventional nano hybrid flowable composite
  Arms: Nanohybrid resin composite

SUMMARY:
The goal of this study is to evaluate the clinical, radiographic and periodontal performance of bioactive Giomer Shofu Flow Plus X F03 compared to nanohybrid resin composite restoration in deep subgingival proximal cavities over a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (20-50)
* Good oral hygiene (plaque index 0 or 1 )
* Patient approving to participate in the study
* Absence of parafunctional habits and/or bruxism

Exclusion Criteria:

* Patients with known allergic or adverse reaction to the tested materials.
* Systematic disease that may affect participation.
* Xerostomic patients.
* Bad oral hygiene (plaque index 2 or 3 )
* Heavy smokers
* Patients undergoing or will start orthodontic treatment
* Patients with removable prothesis

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Recurrent caries | 1 week, 6 months and 12 months
  * Yes: no evidence of caries continuous along the margin
  * No: caries evident continuous with the margin of restoration

SECONDARY OUTCOMES:
Post-operative sensitivity | 1 week, 6 months and 12 months
  * No: Absent
  * Yes: Present
Fracture of the restoration | 1 week, 6 months and 12 months
  * Restoration is intact and fully retained.
  * Restoration is partially retained with some portion of the restoration still intact.
  * Restoration is completely missing
Bleeding on probing | 1 week, 6 months and 12 months
  * 0 Healthy gums
  * 1 Bleeding on probing
  * 2 periodontal problem with bone loss

IPD SHARING:
Plan to Share IPD: Undecided